CLINICAL TRIAL: NCT00038662
Title: A Phase 2 Study Evaluating the Safety and Efficacy of Atrasentan (ABT-627) in Men With Hormone Naive Prostate Cancer Exhibiting Early Signs of Biochemical Failure
Brief Title: Safety and Efficacy of Atrasentan in Men With Hormone Naive Prostate Cancer Exhibiting Early Signs of Biochemical Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01-366; NCT00084994 (obsolete NCT alias)
Record Dates: First submitted 2002-06-03; First posted 2002-06-04 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atrasentan

INTERVENTIONS:
Drug: Atrasentan

SUMMARY:
The purpose of this phase II, randomized, double-blind placebo controlled, multi-center study is to evaluate the safety and efficacy of 10 mg atrasentan in hormone naive subjects as measured by rate of rise in the PSA (primary objective).

ELIGIBILITY:
Inclusion Criteria:

* prostate adenocarcinoma,
* radical prostatectomy,
* PSA between 0.4 and 5 ng/mL,
* PSADT < 1 year

Exclusion Criteria:

* previous hormonal therapy,
* salvage therapy to the pelvis within 3 months prior to randomization

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-05

PRIMARY OUTCOMES:
Evaluate the safety and efficacy of 10mg atrasentan in hormone naive subjects, as measured by the rate of rise in PSA.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Sleep, M.D., Study Director — Abbott
Locations (40):
- United States (24):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Arkansas Urologial Associates, PA, Little Rock, Arkansas
  - San Diego Urology Center, La Mesa, California
  - Western Clinical Research Inc, Torrance, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Clinical Physiology Associates, Fort Myers, Florida
  - Southeastern Urological Center, PA, Tallahassee, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Sheldon Freedman MD, Las Vegas, Nevada
  - VA Medical Center(111), Reno, Nevada
  - Nevada Urology Associates, Reno, Nevada
  - Carolinas Medical Centre, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Urologic Specialists Of Oklahoma, Inc., Tulsa, Oklahoma
  - Oregon Urology Specialists, Eugene, Oregon
  - Urological Assoc. of Lancaster, Lancaster, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Center for Urologic Care, West Reading, Pennsylvania
  - Ntouch Research Corporation, Dallas, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Jeffrey Frankel, M.D., Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Canada (16):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cal Andreou, MD, Surrey, British Columbia
  - Can-Med Medical Research Inc, Victoria, British Columbia
  - Bruce W. Palmer Urology Inc., Kentville, Nova Scotia
  - The Male Health Centres, Barrie, Ontario
  - Burlington Professional Centre, Burlington, Ontario
  - Hamilton & District Urology Association, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Quest Clinical Trials, Markham, Ontario
  - Guardian Medical Arts Bldg., North Bay, Ontario
  - Jack Barkin, MD, North York, Ontario
  - The Male Health Centres, Oakville, Ontario
  - Sunnybrook &Women's College Health Sciens Center, Toronto, Ontario
  - Hopital Notre-Dame, Montreal, Quebec
  - Chuq Pavillon Hotel-Dieu, Québec, Quebec